CLINICAL TRIAL: NCT06365710
Title: A Randomized Controlled Trial Comparing Traditional Physiotherapy vs Telerehabilitation After Volar Plating of Distal Radius Fracture: a Study Protocol
Brief Title: Physiotherapy vs Telerehabilitation After Volar Plating of Distal Radius Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Töölö Hospital (Other)
Responsible Party: Principal Investigator, Samuli Aspinen, Principal investigator, Hospital District of Helsinki and Uusimaa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/206/2022
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Orthopedic Procedures; Physical Therapy Modalities; Postoperative Care; Rehabilitation; Wrist Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): The telerehabilitation group will start the physiotherapy guided by the digital care pathway postoperatively. The pathway includes videos, photos, animations and written material for rehabilitation of the operated hand. The same weightbearing instructions and mobilization exercises are shown in the videos and photos as are instructed in the physiotherapist appointment in the traditional physiotherapy group.
  Interventions: Other: Telerehabilitation
- Traditional Physiotherapy (Active Comparator): The traditional physiotherapy group will attend appointment with the physiotherapist at two-week and five week timepoints. After this, this group can attend additional physiotherapist appointments if seen necessary by the physiotherapist or the surgeon.
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Telerehabilitation — Telerehabilitation program
  Arms: Telerehabilitation
Other: Traditional physiotherapy — Guided rehabilitation program with physiotherapist appointments
  Arms: Traditional Physiotherapy

SUMMARY:
Trial purpose is to research the outcome comparing traditional physiotherapy vs telerehabilitation after volar plating of distal radius fracture.

Patients with distal radius fracture that meet the operative criteria set by the Finnish Current Care guidelines are randomized (1:1 computer generated sequence with random block size) to two parallel groups and will undergo operative treatment and traditional physiotherapy vs telerehabilitation.

Baseline data is collected preoperatively and patients are followed at 1, 3 and 12 months after enrollment. The primary end-point is 3 months and the primary outcome is the Patient-Rated Wrist Evaluation (PRWE).

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture, which applies the surgical requirements
* age between 18 to 65 years
* Non concomitant injuries including ligament injuries and distal ulna fractures, however ulnar styloid avulsion is accepted
* No significant comorbidities
* No previous problems with the examined hand
* Ability to understand Finnish fluently

Exclusion Criteria:

* High energy or multiple injuries
* Open fractures
* Injury of both upper extremities
* Other operative injury on the same side
* Rheumatoid arthritis of other inflammatory joint disease
* Heavy smoker (over 20 cigarettes per day)
* Disease of medication slowing ossification
* Alcohol or drug abuse
* Psychiatric disorder with poor treatment balance
* Neurological disorder which affects the function of the injured extremity
* Fixation material other than a volar locking plate
* Fracture fixation is not stable enough to start rehabilitation after 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) | 12 months
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists two subscales: Pain and Function (0=best possible outcome, 10=worst possible outcome)

SECONDARY OUTCOMES:
Grip strength | 12 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side
Quick Disabilities of the arm, shoulder, and hand | 12 months
  The QuickDASH is self-reported questionnaire and shortened version of DASH outcome measure to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb in 11 dimensions in 1-5 scale (1=best possible outcome, 5=worst possible outcome)
Pain (Visual Analogue Scale) | 12 months
  The VAS is derived by health care professional question of pain in scale 0 to 10 (0=no pain, 10=worst possible pain).
Wrist range of motion (ROM) | 12 months
  Wrist ROM is measured on both wrists with a handheld goniometer in degrees.
Adverse events | 12 months
  Incidence of adverse events (i.e. non-union, fracture, reoperation, infection, iatrogenic tendon/nerve/arterial injury, complex regional pain syndrome, traumatic arthritis) is recorded and compared between study groups.
Global improvement | 12 months
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better
Patient-rated Quality of Life (EQ-5D) | 12 months
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The options are in 5-step scale. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Cost-utility analysis | 12 months
  Quality-adjusted life years/months measured as a change in EQ-5D

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Musculosceletal and Plastic Surgery, Hand Surgery Unit, Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
Public access to the final trial dataset will be available on reasonable request from the principal investigator for research purposes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10 years
Access Criteria: Public access to the final trial dataset will be available on reasonable request from the principal investigator for research purposes. Study protocol, SAP and ICF will be pupblished as a part of the study protocol